CLINICAL TRIAL: NCT07393243
Title: Does Clear Priming of the Cardiopulmonary Bypass Circuit Reduce Bypass Associated Inflammation in Ventricular Septal Defect Patients?
Brief Title: Bypass Clear Priming VSD Cardiopulmonary Bypass Circuit Reduce Bypass Associated Inflammation?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Vishal Nigam, Attending Physician, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003941
Record Dates: First submitted 2024-04-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Septal Defect
Keywords: cardiac surgery; cardiopulmonary bypass; inflammation; blood product
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood prime (No Intervention): The research participants in this arm will undergo their clinically indicated cardiac surgery. The control group will have the bypass pumped primed with mixture of crystalloid solution and blood, which is currently standard of care.
- Clear prime (Experimental): The research participants in this arm will undergo their clinically indicated cardiac surgery. The experimental group will have the bypass pump primed with mixture of crystalloid solution, non-blood fluids.
  Interventions: Procedure: Clear priming of the bypass pump

INTERVENTIONS:
Procedure: Clear priming of the bypass pump — The intervention is priming the pump with non-blood products.
  Arms: Clear prime

SUMMARY:
The purpose of this trial is to study if priming the pump used during cardiac surgery with non-blood fluids instead of donated blood products reduces the inflammation that occurs after heart surgery. The study will focused on pediatric participants who require open heart surgery to repair certain types holes in the heart.

Typically for pediatric patients, the cardiopulmonary bypass pump is "primed" (filled) with donated blood products. This project is going to test if the exposure to these blood products causes inflammation. Patients experience significant inflammation (swelling) after undergoing cardiopulmonary bypass. This inflammation can interfere and slow down the patient's recovery from cardiac surgery. With this project, the investigator are studying if filling the bypass pump with non-blood products reduces the bypass-associated inflammation.

The investigators are also studying if using non-blood fluids to fill the bypass pump reduces bypass associated side effects.

The investigators are also trying to understand how the inflammation starts. The investigators also want to study genetic material called DNA that is collected from a person's blood. Instructions for the body are contained in parts of DNA called genes. Genes determine things like hair and eye color. The investigator hope by studying genes the investigator can learn more about the inflammation that occurs after heart surgery, but the investigators might use participant's genetic information to study other diseases or conditions other the inflammation that occurs after heart surgery.

The investigators will be studying the recovery of 60 participants between 1 month to 18 months of age who require open heart surgery to repair ventricular septal defects (VSDs), a congenital heart defect where there a hole between the lower chambers of the heart.

Participants will:

Allow for information about how the participants recover from surgery to be collected.

Allow blood samples during and after surgery to be collected to understand how the markers of inflammation change between the two groups (blood versus non-blood priming).

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is required for surgical correction/palliation of congenital heart defects. Exposure to CPB results in a robust activation of inflammatory responses. It is now well established that exposure to the CPB circuit is associated with an overwhelming, detrimental systemic inflammatory response. The factors associated with this response may be related to the circuit and exposure to the circuit surface, or may be associated with the body's response to surgical trauma, changes in temperature, etc. Multiple pathways have been shown to be mediating this response, including complement activation, leukocyte activation, endotoxin release, release of oxygen-free radicals, nitric oxide, cytokines, platelet-activation factor, arachidonic acid metabolites and endothelins. Activation of these inflammatory pathways has been implicated in the development of some of the major postoperative complications, such as bleeding tendencies, respiratory insufficiency, renal dysfunction, abnormalities in liver function, and, most seriously, multi-organ failure. Multiple pharmacological therapies have been investigated, with a single aim, to modulate this systemic inflammation. The most widely investigated ones have been corticosteroid administration, use of heparin-coated circuits, leukocyte depletion and ultrafiltration. Despite these efforts, the activation of inflammatory pathways in response to CPB remains a significant clinical problem especially in neonates undergoing CPB.

Over the last several years, several centers including Seattle Children's have been pursuing efforts to restrict the administration of blood products during CPB. In some of the recent publications on the topic, the justifications for moving towards "bloodless CPB" include reducing potential infection risks, consideration that blood products are valuable limited resource, and the concerns of certain religious communities. A limitation of these studies is that they do not examine a patient's clinical course or markers of inflammation in depth. CPB patients experience significant post-CPB inflammation - including increased cytokine levels, inflammatory cell infiltration, vascular leak, and multi-organ dysfunction. In children recovering from complicated cardiac surgeries, increased cytokine levels are associated with high mortality and extended intensive care stays. Typically, a blood-containing prime has been used as a method to preserve high hematocrit levels and maintain oxygen delivery. There are several mechanisms by which exposure to blood products can activate inflammation-which include allergic reactions, cytokines in the blood products, or release of proinflammatory proteins from red blood cells. These mechanisms serve as the basis for the hypothesis that "clear prime" CPB patients will have reduced inflammation as compared to standard of care CPB patients.

Since 5/2021, 174 CPB patients have been operated on at Seattle Children's Hospital (SCH) using restrictive blood management. In 90 of these patients, "bloodless" surgery was attempted. These patients received CPB priming with crystalloid fluids only and without any addition of blood products. These crystalloid fluids are same ones used in current standard of care treatment for pediatric cardiac surgery cases. All other aspects of the patients' treatment were the same including the same bypass machines and tubing. 47 of these patients did not receive blood products during the surgery. 35 patients did not receive any blood products during the hospitalization. There were no statistical differences between the median ventilation time and Intensive Care Unit (ICU) length of stay between the patients operated on with such restrictive blood management as compared to patient controls from our center in which blood products were added to CPB prime.

Dr. Bohuta's recent observational study of 99 SCH neonatal cardiac cases using historical controls identified no statistical difference in postoperative seizures, bleeding events, and lactate levels during CPB between patients who received clear prime versus those who received a blood prime. In this same study, both length of stay and postoperative mechanical ventilation time was shorter in the clear prime group. Hematocrit was consistently lower post-operatively for patients in the crystalloid only group, otherwise, there were no unintended consequences/ adverse events identified in the crystalloid only cohort.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 5-10kg
* Age 1-18 months
* Requiring cardiopulmonary bypass as part of clinically indicated surgery
* Surgery performed by Dr. Bohuta or Dr. Greene

Exclusion Criteria:

* Hemoglobin/hematocrit too low for clear CPB prime (post-dilution Hct <24%)
* Pre-operative ECMO support
* Active infection
* Not clinically appropriate for clear prime (instability, arrhythmias, desaturation, etc.)
* Genetic syndrome
* Pork allergy or family requests pork avoidance

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Changes in RNA expression of the inflammatory marker TNF-α fold pre-cardiopulmonary bypass (CPB) to 24 hours post-CPB | Up to 24 hours post surgery
  Plasma from blood samples collected during four timepoints spanning from pre-CPB to 24 hours post-CPB will be analyzed via RNA-Seq to assess changes in TNF-α fold levels. RNA-Seq measures change in gene expression relative to baseline, with higher relative gene expression indicated higher inflammation.
Changes in protein expression of the inflammatory marker TNF-α fold pre-cardiopulmonary bypass (CPB) to 24 hours post-CPB | Up to 24 hours post surgery
  Plasma from blood samples collected during four timepoints spanning from pre-CPB to 24 hours post-CPB will be analyzed ELISA to assess changes in TNF-α fold levels. ELISA measures concentration in picograms per milliliter, with higher scores indicating more inflammation.
Changes in RNA expression of the inflammatory marker IL8 fold pre-cardiopulmonary bypass (CPB) to 24 hours post-CPB | Up to 24 hours post surgery
  Plasma from blood samples collected during four timepoints spanning from pre-CPB to 24 hours post-CPB will be analyzed via RNA-Seq to assess changes in IL8 fold levels. RNA-Seq measures change in gene expression relative to baseline, with higher relative gene expression indicated higher inflammation.
Changes in protein expression of the inflammatory marker IL8 fold pre-cardiopulmonary bypass (CPB) to 24 hours post-CPB | Up to 24 hours post surgery
  Plasma from blood samples collected during four timepoints spanning from pre-CPB to 24 hours post-CPB will be analyzed via ELISA to assess changes in IL8 fold levels. ELISA measures concentration in picograms per milliliter, with higher scores indicating more inflammation.

SECONDARY OUTCOMES:
Time to extubation | From intubation until extubation (up to 24 hours post-surgery)
  Clinical data will be collected to measure the number of hours and minutes post-surgery until participants are extubated.
Peak lactic acid levels over the first 24 hours post-surgery | Up to 24 hours post-surgery
  Clinical laboratory data will be reviewed to identify the highest lactic acid (Normal: ≤2 mmol/L) value recorded within the first 24 hours after surgery. Lactic acid levels (measured in mmol/L) indicate how well the body is delivering oxygen to tissues after surgery.
Vasoactive-inotropic score over the first 24 hours post-surgery | Up to 24 hours post-surgery
  Clinical data will be collected to determine how much ionotropic support is needed during the first 24 hours after surgery. The vasoactive-inotropic score typically range from 0 to 15, with higher scores indicating a greater need for inotropic support and worse outcomes, and values above 15 are considered atypical.
Length of hospital stay post-surgery | From the date of surgery until the date of hospital discharge, assessed up to 90 days post-surgery.
  Clinical information will be collected from participants' medical charts to measure the length of hospital stay (in days) after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Nigam, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie results in publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication, deidentified IPD will be shared.

REFERENCES:
- [Background] Van Gassen S, Callebaut B, Van Helden MJ, Lambrecht BN, Demeester P, Dhaene T, Saeys Y. FlowSOM: Using self-organizing maps for visualization and interpretation of cytometry data. Cytometry A. 2015 Jul;87(7):636-45. doi: 10.1002/cyto.a.22625. Epub 2015 Jan 8. PMID 25573116
- [Background] Nellis ME, Karam O, Valentine SL, Bateman ST, Remy KE, Lacroix J, Cholette JM, Bembea MM, Russell RT, Steiner ME, Goobie SM, Tucci M, Stricker PA, Stanworth SJ, Delaney M, Lieberman L, Muszynski JA, Bauer DF, Steffen K, Nishijima D, Ibla J, Emani S, Vogel AM, Haas T, Goel R, Crighton G, Delgado D, Demetres M, Parker RI; Pediatric Critical Care Transfusion and Anemia EXpertise Initiative-Control/Avoidance of Bleeding (TAXI-CAB), in collaboration with the Pediatric Critical Care Blood Research Network (BloodNet), and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Executive Summary of Recommendations and Expert Consensus for Plasma and Platelet Transfusion Practice in Critically Ill Children: From the Transfusion and Anemia EXpertise Initiative-Control/Avoidance of Bleeding (TAXI-CAB). Pediatr Crit Care Med. 2022 Jan 1;23(1):34-51. doi: 10.1097/PCC.0000000000002851. PMID 34989711
- [Background] Burnside JL, Ratliff TM, Kelly MN, Naguib AN, Galantowicz M, Hodge A. Bloodless Arterial Switch Operation in a 2.7-kg Jehovah's Witness Patient. J Extra Corpor Technol. 2020 Jun;52(2):142-145. doi: 10.1182/ject-2000003. PMID 32669741
- [Background] Wloch A, Boettcher W, Sinzobahamvya N, Cho MY, Redlin M, Dahnert I, Photiadis J. Bloodless priming of the cardiopulmonary bypass circuit: determinants of successful transfusion-free operation in neonates and infants with a maximum body weight of 7 kg. Cardiol Young. 2018 Oct;28(10):1141-1147. doi: 10.1017/S1047951118001154. Epub 2018 Jul 23. PMID 30033907
- [Background] Faraoni D, Meier J, New HV, Van der Linden PJ, Hunt BJ. Patient Blood Management for Neonates and Children Undergoing Cardiac Surgery: 2019 NATA Guidelines. J Cardiothorac Vasc Anesth. 2019 Dec;33(12):3249-3263. doi: 10.1053/j.jvca.2019.03.036. Epub 2019 Mar 20. PMID 31076306
- [Background] Wypij D, Jonas RA, Bellinger DC, Del Nido PJ, Mayer JE Jr, Bacha EA, Forbess JM, Pigula F, Laussen PC, Newburger JW. The effect of hematocrit during hypothermic cardiopulmonary bypass in infant heart surgery: results from the combined Boston hematocrit trials. J Thorac Cardiovasc Surg. 2008 Feb;135(2):355-60. doi: 10.1016/j.jtcvs.2007.03.067. PMID 18242268
- [Background] Tu LN, Hsieh L, Kajimoto M, Charette K, Kibiryeva N, Forero A, Hampson S, Marshall JA, O'Brien J, Scatena M, Portman MA, Savan R, Benner C, Aliseda A, Nuri M, Bittel D, Pastuszko P, Nigam V. Shear stress associated with cardiopulmonary bypass induces expression of inflammatory cytokines and necroptosis in monocytes. JCI Insight. 2021 Jan 11;6(1):e141341. doi: 10.1172/jci.insight.141341. PMID 33232305
- [Background] Lam LKM, Murphy S, Kokkinaki D, Venosa A, Sherrill-Mix S, Casu C, Rivella S, Weiner A, Park J, Shin S, Vaughan AE, Hahn BH, Odom John AR, Meyer NJ, Hunter CA, Worthen GS, Mangalmurti NS. DNA binding to TLR9 expressed by red blood cells promotes innate immune activation and anemia. Sci Transl Med. 2021 Oct 20;13(616):eabj1008. doi: 10.1126/scitranslmed.abj1008. Epub 2021 Oct 20. PMID 34669439
- [Background] Bohuta L, Charette K, Chan T, Joffe D, Koth A, Greene CL, Mauchley D, McMullan DM. Encouraging results of blood conservation in neonatal open-heart surgery. J Thorac Cardiovasc Surg. 2024 Mar;167(3):1154-1163. doi: 10.1016/j.jtcvs.2023.07.032. Epub 2023 Jul 29. PMID 37517580
- [Background] Bozza MT, Jeney V. Pro-inflammatory Actions of Heme and Other Hemoglobin-Derived DAMPs. Front Immunol. 2020 Jun 30;11:1323. doi: 10.3389/fimmu.2020.01323. eCollection 2020. PMID 32695110
- [Background] Appachi E, Mossad E, Mee RB, Bokesch P. Perioperative serum interleukins in neonates with hypoplastic left-heart syndrome and transposition of the great arteries. J Cardiothorac Vasc Anesth. 2007 Apr;21(2):184-90. doi: 10.1053/j.jvca.2006.02.027. Epub 2006 May 30. PMID 17418729
- [Background] Kato H, Chasovskyi K, Gandhi SK. Are Blood Products Routinely Required in Pediatric Heart Surgery? Pediatr Cardiol. 2020 Jun;41(5):932-938. doi: 10.1007/s00246-020-02338-7. Epub 2020 Mar 13. PMID 32170329
- [Background] Boettcher W, Sinzobahamvya N, Miera O, Redlin M, Dehmel F, Cho MY, Murin P, Berger F, Photiadis J. Routine Application of Bloodless Priming in Neonatal Cardiopulmonary Bypass: A 3-Year Experience. Pediatr Cardiol. 2017 Apr;38(4):807-812. doi: 10.1007/s00246-017-1585-x. Epub 2017 Feb 14. PMID 28197644
- [Background] Naguib AN, Winch PD, Tobias JD, Simsic J, Hersey D, Nicol K, Preston T, Gomez D, McConnell P, Galantowicz M. A single-center strategy to minimize blood transfusion in neonates and children undergoing cardiac surgery. Paediatr Anaesth. 2015 May;25(5):477-86. doi: 10.1111/pan.12604. Epub 2015 Jan 12. PMID 25581204
- [Background] Klein HG. Immunomodulatory aspects of transfusion: a once and future risk? Anesthesiology. 1999 Sep;91(3):861-5. doi: 10.1097/00000542-199909000-00040. No abstract available. PMID 10485799
- [Background] Mou SS, Giroir BP, Molitor-Kirsch EA, Leonard SR, Nikaidoh H, Nizzi F, Town DA, Roy LC, Scott W, Stromberg D. Fresh whole blood versus reconstituted blood for pump priming in heart surgery in infants. N Engl J Med. 2004 Oct 14;351(16):1635-44. doi: 10.1056/NEJMoa041065. PMID 15483282
- [Background] Holmes JH 4th, Connolly NC, Paull DL, Hill ME, Guyton SW, Ziegler SF, Hall RA. Magnitude of the inflammatory response to cardiopulmonary bypass and its relation to adverse clinical outcomes. Inflamm Res. 2002 Dec;51(12):579-86. doi: 10.1007/pl00012432. PMID 12558191